CLINICAL TRIAL: NCT05599230
Title: Daily Monitoring of Respiratory Symptoms and Spirometry During ETI Treatment in Persons With Cystic Fibrosis.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CHC Montlegia (Other)
Responsible Party: Principal Investigator, Lebecque Patrick, Principal investigator, Clinical Professor, CHC Montlegia
Other Study IDs: ML001
Record Dates: First submitted 2022-10-21; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Cystic Fibrosis
Keywords: elexacaftor; time course; FEV1; Respiratory symptoms
MeSH Terms: conditions — Cystic Fibrosis; Signs and Symptoms, Respiratory | interventions — elexacaftor; ivacaftor; tezacaftor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- CF patients before (3 days) and during (14 days) ETI treatment: Patients over 12 years old and eligible will start ETI treatment ( current standart treatment).
  * Morning: Elexacaftor 100 mg, Tezacaftor 50 mg, Ivacaftor 75 mg, 2 tablets
  * Evening: Ivacaftor 150 mg
  Interventions: Drug: Elexacaftor 100 MG / Ivacaftor 75 MG / Tezacaftor 50 MG, 2 tablets each morning + Ivacaftor 150 mg one tablet each evening

INTERVENTIONS:
Drug: Elexacaftor 100 MG / Ivacaftor 75 MG / Tezacaftor 50 MG, 2 tablets each morning + Ivacaftor 150 mg one tablet each evening — Patients will daily perform home spirometry and complete a respiratory symptoms score before (3 days) and during (first 14 days) ETI treatment.

SUMMARY:
The goal of this observational study is to provide optimal monitoring and support when initiating ETI treatment in eligible persons with cystic fibrosis (aged 12 y +) and to document on a daily basis, from 72 hours before the start of treatment and then for 14 days i) i) FEV1 changes (home spirometry), ii) ii) respiratory symptoms changes, iii) any possible side effects. Through a dedicated electronic platform, these data will be monitored every day by the medical team, which will be fully available for any questions or concerns patients may have.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis diagnosis
* At least 12 years old
* Carrier of at least one copy of F508del mutation
* Ability to perform reliable and reproducible spirometry
* Medical and psychological stability
* written consent
* owning a smartphone

Exclusion Criteria:

* Lung transplant
* FEV1 > 120 % pr (%GLI) at the inclusion test
* Pulmonary exacerbation

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: CF patients aged 12 y or more, carrying at least one copy of F508del mutation, in stable condition, reliably performing spirometry
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
FEV1 changes from baseline (3 days before treatment) to Day 14 under ETI | 17 days
  Daily home spirometry with Spirobank device, between 14H-20H, before nebulization and / or physiotherapy

SECONDARY OUTCOMES:
Respiratory symptoms score changes from baseline (3 days before treatment) to Day 14 under ETI | 17 days
  Daily scoring unsing a respiratory questionnaire (8 questions); each item is scored 1 to 5 (worse score: 40)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Lebecque, PhD, Principal Investigator — CHC Montlegia
Locations (1):
- Lebecque, Liège, Belgium